CLINICAL TRIAL: NCT03749356
Title: Multi Center, Non-comparative, Phase IV Study to Evaluate the Efficacy and Safety of Once-Daily Prolonged Release Tacrolimus Capsule(TacroBell SR Cap.) in Kidney Transplant Recipients
Brief Title: Study to Evaluate the Efficacy and Safety of Once-Daily Tacrolimus in Kidney Transplant Recipients
Acronym: OPIRUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211KT18008
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Once-Daily Tacrolimus (Experimental): One arm: TacroBell SR Cap.
  Interventions: Drug: TacroBell SR cap.

INTERVENTIONS:
Drug: TacroBell SR cap. — * Orally, once-daily in the morning
  * After first dose 0.2mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 3~12ng/ml for 0 to 3months and then at 3~8ng/ml for 3 to 6months of study treatment.
  Other Names: Tacrolimus SR cap.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety and of Once-Daily Tacrolimus (TacroBell SR Cap.) in patients who received renal transplantation.

DETAILED DESCRIPTION:
This study is a multi-center, non-comparative, and phase IV clinical trial that evaluates the efficacy and safety of combined Once-Daily Tacrolimus (TacroBell SR Cap.) administration for 24 weeks in patients with immunosuppressive therapies after renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old(male or female)
* Patients who are planning to receive a kidney from a deceased or a living non-related/related donor
* Agreement with written informed consent

Exclusion Criteria:

* Previously received organs other than kidneys or who are planed to be transplanted simultaneously
* Receive a kidney from a donor whose ABO blood type is not compatible with that of the recipient
* Receive a kidney from a related donor who showed HLA-0 mismatch (identical)
* Undergo desensitization therapy with high sensitization
* Diagnosed with cancer in the last five years [Patients, however, who have recovered from skin cancer (squamous cell/basal cell carcinoma) or thyroid cancer can be enrolled.]
* Patients or donors who have positive HIV test result
* Inadequate for registration under the judgment of the investigator due to severe gastrointestinal disorders
* Severe systemic infection requiring treatment
* Prior to the kidney transplantation

  * Treatment with active liver disease or Liver function test(T-bilirubin, AST, ALT)is over 3 times than upper normal limit
  * WBC< 2,500/mm^3, or platelet < 75,000/mm^3, or ANC < 1,300/mm^3
* Pregnant women or nursing mothers
* Fertile women who not practice contraception with appropriate methods
* Participated in other trial within 4 weeks
* In investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure (biopsy-confirmed acute rejection; TCMR, graft loss, death, or follow-up failure) | until 24 weeks
  The frequency and percentage of composite efficacy failure(biopsy-confirmed acute rejection; TCMR, graft loss, death, or follow-up failure)

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection(TCMR, AMR) | until 24 weeks
  The frequency and Incidence
Pathological results of acute rejection | until 24 weeks
  By Banff classification categories
Survival rate of transplated organ | at 24 weeks
  Kaplan-Meier
Survival rate of Patients | at 24 weeks
  Kaplan-Meier
Serum-Cr, eGFR | at 24 weeks
  eGFR using CKD-epi method
Evaluate safety of TacroBell SR. cap. from number of participants with adverse events | until 24 weeks
  safety data

CONTACTS AND LOCATIONS:
Overall Officials: Yu Seun Kim, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea